CLINICAL TRIAL: NCT00518479
Title: Pathophysiological Mechanisms of Hypertensive LVH:Optimising Regression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr JP Greenwood, Senior Lecturer, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG/03/001
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
Keywords: Hypertension; Left Ventricular Hypertrophy
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Bendroflumethiazide; Amlodipine; Valsartan; moxonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Neurohormonal stimulatory arm
  Interventions: Drug: Bendroflumethiazide 2.5mg OD; Amlodipine 10mg OD
- 2 (Experimental): Neurohormonal inhibitory arm
  Interventions: Drug: Valsartan 160mg OD; Moxonidine 400mcg OD

INTERVENTIONS:
Drug: Bendroflumethiazide 2.5mg OD; Amlodipine 10mg OD
  Arms: 1
Drug: Valsartan 160mg OD; Moxonidine 400mcg OD
  Arms: 2

SUMMARY:
Uncontrolled high blood pressure can cause heart muscle 'thickening', and this increases the likelihood of complications and death. The high blood pressure explains some but not all of this increase in heart size. This study will investigate the other causes, and will measure the heart muscle 'thickness' very accurately using the latest and most accurate technique called cardiac magnetic resonance imaging (MRI). The best way to treat this heart thickening remains to be determined. We hope to be able to show that by specifically targeting the cause of heart muscle thickening we can reduce its occurrence more effectively than by other standard means of blood pressure treatment

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed essential hypertension (within 6 months).
* Age 25 to 80 years; Weight < 100kg.
* Sinus rhythm without significant ventricular or atrial ectopy.

Exclusion Criteria:

* Current angiotensin II receptor antagonist or ACE Inhibitor treatment.
* Contra-indication to any of the protocol anti-hypertensive agents.
* Angina requiring treatment with a Beta blocker or calcium antagonist
* Any disease affecting the autonomic nervous system e.g. congestive cardiac failure, diabetes, neurological disease, malignancy, pregnancy.
* Contraindication to MRI (pacemaker, intra-orbital debris, intra-auricular implants, intra-cranial clips, history of claustrophobia, inability to lie supine for 15 minutes etc).

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-09; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is decrease in LV mass as assessed by cardiac MRI compared between the two treatment groups. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John P Greenwood, MBChB, PhD, Principal Investigator — Leeds University
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, Wesst Yorkshire, United Kingdom

REFERENCES:
- [Result] Burns J, Sivananthan MU, Ball SG, Mackintosh AF, Mary DA, Greenwood JP. Relationship between central sympathetic drive and magnetic resonance imaging-determined left ventricular mass in essential hypertension. Circulation. 2007 Apr 17;115(15):1999-2005. doi: 10.1161/CIRCULATIONAHA.106.668863. Epub 2007 Mar 26. PMID 17389264